CLINICAL TRIAL: NCT04914338
Title: Feasibility of a Multidisciplinary Approach to Circumvent Healthspan Decline After Allogeneic Hematopoietic Cell Transplantation in Older Patients
Brief Title: A Multidisciplinary Approach to Improve the Health of Older Adults With Blood Cancers After Stem Cell Transplantation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21026; NCI-2021-03939 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21026 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2021-05-24; First posted 2021-06-04 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Health Promotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive care (MDT-intervention) (Experimental): Patients participate in the MDT-intervention including access to a HCT physician, a geriatrician, physical or occupational therapist, dietician, and a social worker for three months before HCT and up to 100 days after HCT.
  Interventions: Other: Health Promotion; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Health Promotion — Participate in MDT-intervention
  Other Names: Health Promotion (Salutogenesis); Health Promotion and Wellness; Mindfulness Health Promotion; Salutogenesis
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies the usefulness and process of a multidisciplinary intervention, where patients see multiple healthcare professionals, aimed at improving fitness and the ability to bounce back after transplant for older adults with blood cancers planned for stem cell transplantation. Using a multidisciplinary team approach may increase patients' ability to withstand the transplant by optimizing health to better prepare patients for the expected complications after stem cell transplantation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the feasibility of delivering a geriatric assessment guided by a multi-disciplinary team (MDT) intervention before allogeneic hematopoietic cell transplantation (HCT) in older patients.

SECONDARY OBJECTIVES:

I. Establish successful dose intensity of resiliency bolstering. II. Describe HCT utilization among enrolled patients. III. Create a standardized and exportable library of MDT-facilitated interventions.

IV. Estimate the benefit derived from the MDT approach compared to historic controls for day +100 outcomes of falls, delirium and functional decline.

V. Quantify early functionally independent survival (FIS) to estimate HCT-associated health span decline.

EXPLORATORY OBJECTIVES:

I. Characterize reasons patients do not undergo HCT after MDT intervention. II. Associate early FIS with 1-year non-relapse mortality (NRM) and overall survival (OS).

III. Integrate virtual assessment and interventions. IV. Correlate image defined sarcopenia with objective function. V. Biobank blood and stool for future studies of accelerated aging.

OUTLINE:

Patients participate in the MDT-intervention including access to a HCT physician, a geriatrician, physical or occupational therapist, dietician, and a social worker for three months before HCT and up to 100 days after HCT.

After completion of study, patients are followed up for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant
* >= 65 years at time of planned HCT infusion
* Anticipated to be candidate for allogeneic transplant per treating physician at the time of enrollment
* Ability to read English, Spanish or Mandarin. Other languages will be acceptable with principal investigator (PI) agreement if surveys are available and language does not preclude completing study procedures
* Any conditioning regimen and allogeneic donor permitted
* Hematologic malignancy or disease as indication for HCT
* Willing and able to complete study requirements

Exclusion Criteria:

* Prior allogeneic stem cell transplant
* Syngeneic donors for HCT
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2026-02-03 (Estimated); Study Completion 2026-02-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of multidisciplinary team (MDT) (met 90 percent threshould, yes / no) | Up to 1 year
  Patients are expected to see 6 providers. Success is defined as enrolled patients seen at least 4 out of six providers. The study will meet feasibility endpoint if 90 percent or more of the enrolled patients are flagged as successful. Each patient will be measured as success or failure according to these rules.

SECONDARY OUTCOMES:
Dose intensity of resiliency bolstering | Up to 1 year
  Adequate dose intensity arbitrarily will be defined as completion of at least 11 of 16 process metrics (i.e, approximately 70 percent of more of process measures).
Rate of hematopoietic cell transplantation (HCT) utilization | Up to 1 year
  Measured by summarizing proportion of patients proceeding to allogeneic HCT.
Library of MDT-facilitated intervention | Up to 1 year
  Will provide a standardized library of evaluation and interventions from the MDT approach. A manual of procedures will be created and a database to capture metrics. Will be categorized by the MDT in a Likert scale to the following question: "Is the library of MDT-facilitated interventions ready to be exposure for a randomized controlled trial".
Functional independent survival (FIS) | Days 30, 60, 100
  FIS will be calculated as with first observed failure events of intensive care unit admissions, delirium, falls, or frail 4 meter walk at day 30 or day 100. Functional impairment will use the milestones of day 30, day 60 day 100.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Artz, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Nedical Center, Duarte, California, United States